CLINICAL TRIAL: NCT02598947
Title: The POST Study; POsterior Shoulder Tightness in Rotator Cuff Related Disorders: A Randomised Controlled Feasibility Study
Brief Title: The POST Study; POsterior Shoulder Tightness in Rotator Cuff Related Disorders
Acronym: POST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sussex Hospitals NHS Trust (Other)
Collaborators: University of Brighton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDRF-2014-05-003
Record Dates: First submitted 2015-10-01; First posted 2015-11-06 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Shoulder Impingement Syndrome
Keywords: posterior shoulder tightness; shoulder impingement syndrome; Glenohumeral joint; exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome; Motor Activity | interventions — Musculoskeletal Manipulations; Exercise; Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior shoulder tightness group (Experimental): As well as receiving a strengthening program for the scapular and rotator cuff musculature, subjects allocated to the 'posterior shoulder tightness' treatment group will also receive specific manual therapy and home stretches to address stiffness of the posterior shoulder
  Interventions: Other: Manual therapy
- Posterior shoulder tightness sham group (Sham Comparator): The 'sham posterior shoulder tightness' group will receive the same strengthening program for the scapular and rotator cuff musculature, in addition they will receive home stretches and manual therapy of similar durations to the 'posterior shoulder tightness' group, but delivered to structures that have no known direct structural influence on the posterior shoulder
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — Exercise, behaviour change interventions and manual therapy
  Other Names: Exercise; Education; Behaviour change interventions

SUMMARY:
Shoulder impingement syndrome is a very common cause of shoulder pain and normally treated with physiotherapy or surgery. Research has shown that physiotherapy is as effective as surgery, however, the incidence of surgery for this condition is on the rise internationally, nationally and locally. The most effective form of physiotherapy, however, is not known. Laboratory studies have suggested that posterior shoulder tightness may contribute to irritation of the soft tissue around the shoulder joint and perpetuate pain from shoulder impingement syndrome. There is a lack of good quality evidence to support this perspective. The aim of this study is to assess the feasibility of conducting a randomized controlled trial to evaluate the effectiveness of treatment for posterior shoulder tightness in combination with 'best care' compared with 'best care' alone in individuals with shoulder impingement syndrome.

The study will be a randomised, controlled, double blind (patient and assessor), parallel group, feasibility study with 1:1 allocation ratio. Patients awaiting surgery will be assessed for inclusion/exclusion criteria and then randomly allocated into one of two groups. 60 patients will be assigned to receive 'best care' physiotherapy, with or without treatment for posterior shoulder tightness.

Physiotherapy treatment will be delivered over 13-15 weeks and outcomes will be assessed at 0, 6-8, 13-15, 26 and 52 weeks. The results will help us to understand if this is an important part of physiotherapy treatment, which might help reduce patient's pain and disability as well as reduce the cost of treatment for the National Health Service.

DETAILED DESCRIPTION:
The study will be a randomised, controlled, double blind (patient and assessor), parallel group, feasibility study with 1:1 allocation ratio. The patients will be assessed for inclusion/exclusion criteria and then randomly allocated into one of two groups. Both groups will receive the same exercise and educational interventions. The treatment group will also receive specific intervention for posterior shoulder tightness; the placebo group will receive placebo posterior shoulder tightness intervention.

Study setting

The study will take place in secondary care environment. Subjects will be recruited from the outpatient orthopaedic clinics at Worthing and Southlands Hospitals, part of Western Sussex Hospitals NHS Foundation Trust.

Recruitment

Recruitment will be promoted with fliers and research posters in the outpatients department. The chief investigator or a research assistant will attend the orthopaedic shoulder clinics and will approach patients in the waiting area to introduce the study and hand out fliers. The orthopaedic team will also introduce the study to patients where appropriate and introduce the patient to the chief investigator or the research assistant if the patient expresses an interest in receiving more information relating to the study.

Where appropriate the chief investigator or the research assistant will ask the patient if they would be willing to be contacted by the chief investigator the following day to discuss the study further. If so the patient details will be passed to the chief investigator who will call the patient at least 24 hours after the introduction of the study. The chief investigator will call to discuss the study further and if the patient is happy to participate an appointment will be arranged for the patient to attend the physiotherapy department of either Worthing or Southlands hospital. At this time informed consent, eligibility assessment and baseline outcome measurement will be performed. In addition baseline characteristics will be recorded in an attempt to minimize selection bias. The estimated time for this visit is 90 minutes.

Randomisation and Blinding

Prior to subject randomisation, sealed envelopes will be prepared containing the treatment manual for the two treatment arms. The assessor will assign consenting participants a unique study number and the anonymised data will be forwarded to the named research officer at the Brighton and Sussex Clinical Trials Unit (B&S CTU). The officer will enter the data into the software package 'sealed envelope' that will process the data and assign the subject to the treatment or placebo group. An E-mail containing group allocation will then be sent to the assessor. The patient will then be transferred to the reception of the physiotherapy department where the appropriately numbered envelop will be placed with the physiotherapy notes and the patient booked for their initial physiotherapy session. The group allocation of each patient will only be available to the treating physiotherapist when the envelope containing the manual is opened at the initial physiotherapy consultation. The physiotherapist will be instructed not to advise the patient to which group they have been allocated.

Data collection

Data collection will take place prior to random allocation, half way through the intervention (6-8 weeks) and at the end of the intervention (13-15 weeks). At 26 and 52 weeks a telephone follow-up interview will repeat collection of Shoulder pain and Disability Index (SPADI) and the EuroQol questionnaire (EQ-5D-5L) and evaluate the surgical outcome. The chief investigator will perform data collection, an assistant will accompany to assist with measurement of posterior shoulder tightness. The assessor will be blind to the group allocation of participants. Where possible the participants will complete questionnaires unassisted, where assistance is required additional explanation will be provided by the research assistant. Physical data will be collected in the form of a clinical examination at baseline, 6-8 weeks and at 13-15 weeks. The examination will involve measurement of posterior shoulder tightness through the use of three clinical tests. These tests will be performed with measurement brace and digital inclinometer. A reliability study of these three clinical tests has been performed by the chief investigator at the University of Brighton following approval by the Faculty of Health Sciences Research Ethics and Governance Committee. The three clinical tests to identify patients with posterior shoulder tightness are; horizontal adduction, internal rotation in 90 degrees abduction and low flexion.

Physiotherapy intervention

The treatment intervention will be delivered in the physiotherapy outpatient departments of Worthing Hospital or Southlands Hospital. Treatment will be delivered by NHS physiotherapists over 13-15 weeks and consist of 6-8 sessions of physiotherapy. The first 4 sessions will be delivered weekly and the subsequent 4 sessions will be delivered every 2 weeks. This treatment dose and duration is consistent with previous high quality studies (Holmgren et al. 2014, Bernhardsson et al. 2011). The intervention will be delivered while patients are on the surgical waiting list for subacromial decompression surgery. The current waiting times for surgery vary considerably between consultants, from 18-28 weeks. This means the intervention can be fully completed during the waiting time for surgery.

All treatment will be provided by NHS physiotherapist as part of their daily caseload. They will be allocated 45 minutes for initial assessment and 30 minutes for subsequent treatment sessions, in line with current departmental procedure. All therapists will be recruited for the trial on a voluntary basis. Appropriate training will be provided to all physiotherapists. It is estimated that 2 physiotherapists from each of the three physiotherapy sites will be required to deliver the physiotherapy interventions.

For both groups, physiotherapy treatment will consist of education regarding the nature of the patients condition, and the prescription of an exercise program to be performed once a day at home. Each group will perform three strengthening exercises to address the muscular systems of the scapular and rotator cuff musculature and a stretching exercise for the anterior shoulder. The exercises have been selected based on review of the available literature relating to muscular dysfunction in shoulder impingement, electromyography (EMG) studies of shoulder exercises and RCTs where the interventions have been adequately described. The exercises with be taught by the physiotherapist and reviewed at each session where the exercises will be progressed or regressed depending on the patients response since the last visit.

In addition subjects allocated to the 'posterior shoulder tightness' treatment group will also receive specific manual therapy during each physiotherapy session. The treatment has been designed to mobilise the structures of the posterior shoulder. They will be prescribed home stretches to address stiffness of the posterior shoulder.

The 'sham posterior shoulder tightness' group will receive home stretches and manual therapy of similar durations to the 'posterior shoulder tightness' group, but delivered to structures that have no known direct structural influence on the posterior shoulder. The intention is for subjects to receive a similar dose of manual therapy to control for the generic effects of manual therapy, which may have pain relieving mechanisms. The sham intervention will be controlled for time and attention in order to create a comparable attention-control group. Using this design it may be possible to determine if there is any additional benefit to treating posterior shoulder tightness in combination with high quality rehabilitation for patients with shoulder impingement syndrome.

All subjects will be asked to perform 4 strengthening exercises each day and 2 stretches each day as well as attending 6-8 physiotherapy treatments over a 13-15 week period. The exercises will take approximately 10-15 minutes to perform.

The study has been designed as a feasibility study as there are believed to be too many unknown factors to proceed directly to definitive randomised controlled study design. These are outlined in full in section 11A. It is predicted recruitment will begin in May 2016 and continue until November 2018. Final follow-up assessment will occur one year after initial outcome assessment. So it is predicted that final patient contact will occur in October/November 2019.

The study design was discussed in depth with a user group at its conception in June 2013 and two patient representatives have continued to assist throughout the study design. Patients have reviewed the recruitment strategy, patient information literature and consent forms. They have agreed to participate in an informed consent rehearsal and appraisal prior to the start of recruitment to ensure informed consent is thorough and easy for the patient to comprehend and allows sufficient time for questions.

The study steering committee will meet every 6 months to ensure the study is running smoothly. The steering committee will include; Kevin Hall (lead researcher), Chris Mercer (Physiotherapy Consultant, physiotherapy clinical lead), Professor Ann Moore (academic supervisor, or a member of the academic supervisory team), Mr Nurang (Orthopaedic Shoulder Consultant), Richard Brunton (service user), Pamela Clarke (service user), Clare Meachin (Research and Innovation Department) and Physiotherapist (to be confirmed).

Progress reports will be submitted to the National Institute of Health Research (NIHR) at 6 months and then annually for the 5 year duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Listed for subacromial decompression surgery by a consultant orthopaedic surgeon
2. Presence of posterior shoulder tightness, based on a positive result in 2 of 3 clinical tests (see below for explanation)
3. Comprehensive in spoken and written English
4. Site of mechanical pain consistent with shoulder impingement syndrome
5. At least 3 months duration of shoulder pain
6. A minimum SPADI score of 20
7. Clinical examination revealing a positive tests for pain with either Neer's test or Hawkins-Kennedy test

Using the SEM values obtained from the recent reliability study conducted at the University of Brighton (see appendix 1), side-to-side differences of more than 2×SEM are associated with a 95% probability that the difference is not caused by the inaccuracy of the clinical test. Using the SEM values obtained from this study, it is possible to be 95% confident that the difference identified is not due to an error of measurement when the side-to-side difference is greater than;

* 7.4 degrees for horizontal adduction
* 9.6 degrees for internal rotation in abduction
* 7 degrees for low flexion

Based on these results a side-to-side difference of 10 degrees or more on two out of three clinical tests will be considered positive for the presence of posterior shoulder tightness.

Clustering tests enables the clinician to overcome the inherent weaknesses of individual tests. Making a decision relating to the presence of posterior shoulder tightness on the outcome of a cluster of tests may better reflect the complex anatomy of the posterior shoulder and the multiple layers of connective tissue and muscle acting as passive restraint to movement.

Exclusion Criteria;

1. Clinically detectable large full thickness rotator cuff tear
2. Recent trauma (last 3 months) involving the shoulder
3. Clinical and radiologically evidence of osteoarthritis of the glenohumeral joint
4. Symptomatic osteoarthritis of the acromioclavicular joint
5. Adhesive capsulitis (50% deficit of range of movement in 2 or more directions)
6. Malignancy
7. Previous fracture or surgery of the symptomatic shoulder
8. Polyarthritis
9. Past diagnosis of fibromyalgia
10. Rheumatiod arthritis
11. Cervical source of shoulder pain; somatic or radicular (reproduction of familiar shoulder pain during a clinical examination of the cervical spine)
12. Ipsilateral shoulder dislocation in last 2 years
13. Multidirectional instability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (Change) | Baseline, 6-8, 13-15, 26 and 52 weeks.
  Questionnaire relating to pain and disability

SECONDARY OUTCOMES:
EQ-5D-5L (Change) | Baseline, 6-8, 13-15, 26 and 52 weeks.
  Health related quality of life questionnaire
Range of motion; glenohumeral internal rotation, low flexion, horizontal adduction (Change). Range will be assessed using purpose built brace (with built in digital inclinometer) and range will be measured in degrees. | Baseline, 6-8, 13-15 weeks
  Measurement of shoulder movements.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, MSc, Principal Investigator — Western Sussex Hospitals NHS Trust
Locations (1):
- Kevin Hall, Shoreham-by-Sea, Sussex, United Kingdom

REFERENCES:
- [Background] Bernhardsson S, Klintberg IH, Wendt GK. Evaluation of an exercise concept focusing on eccentric strength training of the rotator cuff for patients with subacromial impingement syndrome. Clin Rehabil. 2011 Jan;25(1):69-78. doi: 10.1177/0269215510376005. Epub 2010 Aug 16. PMID 20713438
- [Result] Holmgren T, Hallgren HB, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. Br J Sports Med. 2014 Oct;48(19):1456-7. doi: 10.1136/bjsports-2014-e787rep. PMID 25213604